CLINICAL TRIAL: NCT00001976
Title: CMV Real-Time PCR Versus PP65 Antigenemia in Diagnosing Cytomegalovirus Disease in Hematopoietic Stem Cell Transplant Patients
Brief Title: Comparison of Two Test Methods-NASBA and Antigenemia-for Detecting Cytomegalovirus Infection
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000059; 00-I-0059
Record Dates: First submitted 2000-01-20; First posted 2000-01-21 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-02

CONDITIONS: Cytomegalovirus Infection; Infection
Keywords: CMV; Infection; Comparison; Observational; Cytomegalovirus; RT-PCR
MeSH Terms: conditions — Cytomegalovirus Infections; Infections

SUMMARY:
This study will evaluate the reliability of a new test called Real-Time Polymerase chain reaction (RT PCR) in detecting cytomegalovirus (CMV) in the blood and predicting the course of CMV disease in patients who have recently had a bone marrow transplant. The test's effectiveness will be compared with that of the "pp65 antigenemia assay" now routinely used for this purpose.

CMV is a common virus that is transmitted from person to person by close personal contact. In most healthy people, CVM can remain in the body indefinitely without causing any harm. But, in people with weakened immune systems-including those who have just undergone bone marrow transplant-CMV infection can cause serious, and possibly fatal, complications. Drugs are available to treat this infection, however. Optimum treatment depends on early and accurate detection.

Patients aged 10 to 80 years who are scheduled to undergo bone marrow transplant at the NIH Clinical Center as part of an NIH protocol may be eligible for this 2-phase study. In phase 1, patients will have blood drawn for both RT PCR and antigenemia testing once before the bone marrow transplantation and then weekly for the first 100 days after the transplant. During Phase 2-which begins immediately after the end of phase 1 and continues for one year after the transplant-blood samples for both tests will be drawn up to once a week. The samples for both tests will be collected at the same time and will be taken through a catheter (a thin flexible tube inserted into a vein) that has already been placed for the transplant study. RT PCR testing will require an extra 5 milliliters (1 teaspoon) above what is needed for antigenemia testing, amounting to a maximum of about one-half pint extra over the course of the 1-year study.

It is hoped that the new RT PCR test will prove to be more accurate in detecting CMV infection and predicting disease development, thus enabling doctors to plan early and effective treatment.

DETAILED DESCRIPTION:
Currently, it is the standard of care to use the pp65 antigenemia assay to guide anti-cytomegalovirus therapy in hematopoietic stem cell transplant patients. Nevertheless, over the past two years at our institution, only approximately 10% of antigenemia-positive patients went on to develop overt CMV disease and only 22% of patients with documented clinical CMV disease had a positive antigenemia test in the two weeks prior to diagnosis (data on file).

Recently, a test called CMV Real-Time PCR has been applied to the diagnosis of CMV infection. Preliminary data suggests that this test may be of value in detecting active CMV replication. Thus, it may be able to predict CMV disease and help guide antiviral therapy.

We propose a prospective observational study comparing CMV Real-Time PCR test and pp65 antigenemia. This will be done by taking an extra blood sample (approximately 5 mL) for the CMV Real-Time PCR test from hematopoietic stem cell transplant patients whenever a sample for the pp65 antigenemia test is drawn. No separate venipunctures are anticipated. These samples will be drawn on an approximately weekly basis during the first 100 days post-transplant, as is currently done for the pp65 antigenemia test alone. Additionally, at any time blood is drawn for the pp65 antigenemia test after 100 days, we will also take blood for the CMV Real-Time PCR test, up to one year post-transplant. The results of the CMV Real-Time PCR test will not be used to guide therapy. Overt CMV disease will be identified via real-time chart review and patient interviews by one of the investigators in the study. The primary goal of the study is to evaluate the ability of the CMV Real-Time PCR test to accurately detect active CMV viral proliferation and predict ultimate overt CMV disease as compared to the currently-used pp65 antigenemia test.

ELIGIBILITY:
Male or female patients that are 10 years of age or older up to 80 years of age are included.

Patients must be enrolled in a protocol at the NIH Clinical Center that will result in the patient receiving an allogeneic stem cell transplant (A-HSCT).

Patients who have not yet received a pre-transplant chemotherapy and radiation therapy conditioning regimen are eligible.

Patients must not have a negative IgG serologic test for CMV and whose hematopoietic stem cell donor also has a negative IgG serologic test as reported by the Bone Marrow Transplant staff.

Patients must not have documentation of prior cytomegalovirus antigenemia or disease prior to starting the conditioning regimen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180
Dates: Start 2000-01; Study Completion 2003-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Sable CA, Donowitz GR. Infections in bone marrow transplant recipients. Clin Infect Dis. 1994 Mar;18(3):273-81; quiz 282-4. doi: 10.1093/clinids/18.3.273. No abstract available. PMID 8011804
- [Background] Rowe JM, Ciobanu N, Ascensao J, Stadtmauer EA, Weiner RS, Schenkein DP, McGlave P, Lazarus HM. Recommended guidelines for the management of autologous and allogeneic bone marrow transplantation. A report from the Eastern Cooperative Oncology Group (ECOG). Ann Intern Med. 1994 Jan 15;120(2):143-58. doi: 10.7326/0003-4819-120-2-199401150-00008. PMID 8256974
- [Background] Boeckh M, Gooley TA, Myerson D, Cunningham T, Schoch G, Bowden RA. Cytomegalovirus pp65 antigenemia-guided early treatment with ganciclovir versus ganciclovir at engraftment after allogeneic marrow transplantation: a randomized double-blind study. Blood. 1996 Nov 15;88(10):4063-71. PMID 8916975